CLINICAL TRIAL: NCT01127464
Title: A Randomized, Placebo-controlled, Dose-escalating, Double-blinded Phase I Study to Evaluate the Safety and Immunogenicity of Anti-DEC-205 Monoclonal Antibody (Mab) Targeted HIV Gag p24 Vaccine (DCVax-001) With Poly ICLC (Hiltonol) as Adjuvant in HIV-uninfected Healthy Volunteers
Brief Title: DCVax Plus Poly ICLC in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SSC-0710
Record Dates: First submitted 2010-05-19; First posted 2010-05-20 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: HIV-1 Infection; HIV Infection; Healthy Volunteers
Keywords: HIV-1; HIV preventative vaccine; Healthy Volunteers
MeSH Terms: conditions — HIV Infections | interventions — poly ICLC

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- .3 dose level of DCVax -001 (Experimental): .3 dose level of DCVax plus fixed dose of 1.6 ml Poly ICLC
  Interventions: Drug: DCVax-001; Drug: Poly-ICLC
- 1 mg dose level of DCVax -001 (Experimental): 1 mg dose level of DCVax -001 plus 1.6 ml of poly ICLC
  Interventions: Drug: DCVax-001; Drug: Poly-ICLC
- 3 mg dose level of DCVax-001 (Experimental): 3 mg dose level of DCVax-001 plus poly ICLC
  Interventions: Drug: DCVax-001; Drug: Poly-ICLC
- Placebo (Placebo Comparator): sterile saline
  Interventions: Drug: Placebo
- poly-ICLC alone (Experimental): 1.6 mg of poly-ICLC alone
  Interventions: Drug: Poly-ICLC

INTERVENTIONS:
Drug: DCVax-001 — Comparison of 3 different doses of DCVax-001 administered with poly-ICLC, the administration of poly-ICLC alone, or a placebo control
  Arms: .3 dose level of DCVax -001; 1 mg dose level of DCVax -001; 3 mg dose level of DCVax-001
Drug: Poly-ICLC — Comparison of 3 different doses of DCVax-001 administered with poly-ICLC, the administration of poly-ICLC alone, or a placebo control
  Arms: .3 dose level of DCVax -001; 1 mg dose level of DCVax -001; 3 mg dose level of DCVax-001; poly-ICLC alone
Drug: Placebo — Comparison of 3 different doses of DCVax-001 administered with poly-ICLC, the administration of poly-ICLC alone, or a placebo control
  Arms: Placebo

SUMMARY:
DCVax-001 is a recombinant protein vaccine designed to prevent and potentially treat human immunodeficiency virus (HIV) infection. The vaccine is composed of a fusion protein containing a human monoclonal antibody specific for the dendritic cell receptor, DEC-205 (CD205), and the HIV gag p24 protein. The vaccine is designed to target HIV antigens directly to endocytic pathways in dendritic cells (DCs) that allow for efficient processing and presentation of multiple HIV peptides on both MHC class I and II products, which will induce HIV-specific CD8+ and CD4+ T cells. This vaccine candidate must be combined with appropriate immunostimulants (adjuvants) to induce immunity to the antigen. In the proposed clinical trial we will use poly ICLC (Hiltonol) from Oncovir, Inc as the adjuvant.

DETAILED DESCRIPTION:
This trial will investigate whether delivery of HIV antigens via immunization with anti-DEC-205 p24 monoclonal antibody plus poly ICLC, as an adjuvant, is safe and induces either cellular or humoral immunogenicity in healthy volunteers. We propose to assess the quality of immunity elicited by DEC targeted vaccines in humans. Immunogenicity after HIV antigen delivery directly to dendritic cells could provide the proof-of-concept that dendritic cell targeted protein vaccines may serve as a stand-alone vaccine strategy or in combination with other vaccine modalities against HIV or other diseases.

The main hypothesis of this study is to assess the delivery of HIV antigens via immunization with anti-DEC-205 p24 monoclonal antibody (DCVax-001) plus poly ICLC (Hiltonol) is safe and induces either cellular or humoral immunogenicity in HIV-uninfected, healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult males and females, as assessed by a medical history, physical exam, and laboratory tests
2. Age of at least 18 years of age on the day of screening and no greater than 60 years at time of vaccination
3. Willing to comply with the requirements of the protocol and available for follow-up for the planned duration of the study (screening plus 15 months)
4. In the opinion of the principal investigator or designee, has understood the information provided. (Written informed consent needs to be given before any study-related procedures are performed)
5. Amenable to HIV risk reduction counseling, committed to maintaining behavior consistent with low risk of HIV exposure through the last required protocol clinic visit
6. Assessed by the clinic staff as being at "low risk" for HIV infection on the basis of sexual behaviors within the 12 months prior to enrollment defined as follows:

   * Sexually abstinent OR
   * Had two or fewer mutually monogamous relationships with partners believed to be HIV-uninfected and who did not use illicit drugs (illicit drug use or abuse that includes any injection drugs, methamphetamines (crystal meth), heroin, cocaine, including crack cocaine or chronic marijuana abuse) OR
   * Had two or fewer partners believed to be HIV-uninfected and who did not use illicit drugs (as defined above) and with whom he/she regularly used condoms for vaginal and anal intercourse;
7. If sexually active female, using an effective method of contraception (combined oral contraceptive pill; injectable contraceptive; diaphragm; Intra Uterine Device (IUD); condoms; anatomical sterility in self or partner) throughout the study period. All female volunteers must be willing to undergo urine pregnancy tests at time points as indicated
8. If sexually active male, willing to use an effective method of contraception (such as condoms, anatomical sterility) from screening until 4 weeks after last vaccination (same as above) and will be advised not to get his partner(s) pregnant

Exclusion Criteria:

1. Confirmed HIV-1 or HIV-2 infection
2. Any clinically significant abnormality on history or examination including history of immunodeficiency or autoimmune disease; use of systemic corticosteroids immunosuppressive anticancer, or other medications considered significant by the trial physician within the last 6 months
3. Any clinically significant acute or chronic medical condition requiring care of a physician (e.g., diabetes, coronary artery disease, rheumatologic illness, malignancy, substance abuse) that in the opinion of the investigator would preclude participation
4. Any laboratory value outside of reference range, with the exception of any non-clinically significant Grade I elevations of liver function tests (AST, ALT, direct/total bilirubin), electrolytes, CO2, CBC, urinalysis as determined by the Principal Investigator or his designee as well as creatinine if the estimated glomerular filtration rate is > 60 mL/min/1.73 m2
5. Within the 12 months prior to enrollment, the volunteer has had excessive daily alcohol use or frequent binge drinking or chronic marijuana abuse or any other use of illicit drugs
6. Within the 12 months prior to enrollment, the volunteer has a history of newly-acquired syphilis, gonorrhea, non-gonococcal urethritis, herpes simplex virus type 2 (HSV2), Chlamydia, pelvic inflammatory disease (PID), trichomonas, mucopurulent cervicitis, epididymitis, proctitis, lymphogranuloma venereum, chancroid, hepatitis B (surface antigen, HbsAg) or hepatitis C (HCV antibodies)
7. If female, pregnant, planning a pregnancy during the trial period, or lactating
8. Receipt of a live attenuated vaccine within 30 days or other vaccine within 14 days prior to DEC-205 vaccination
9. Receipt of another experimental HIV vaccine at any time
10. Receipt of blood transfusion or blood products 6 months prior to vaccination
11. Participation in another clinical study of an investigational product currently or within past 12 weeks, or expected participation during this study
12. History of severe local or systemic reactogenicity to vaccination or history of severe allergic reactions
13. Major psychiatric illness
14. In the opinion of the investigator, unlikely to comply with protocol

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2010-05; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | 64 weeks
  The proportion of volunteers with moderate local reactogenicity events; Proportion of volunteers with moderate systemic reactogenicity events; Proportion of volunteers with other moderate adverse events; Proportion of volunteers with serious adverse events; Proportion of volunteers with severe and moderate local and systemic reactogenicity events and adverse events.

SECONDARY OUTCOMES:
Immunogenicity | 64 weeks
  The proportion of volunteers with HIV-1 specific T-cell responses as quantified by IFNγ-ELISpot; The proportion of volunteers with HIV-1 specific T-cell responses as quantified by multiparametric cytokine flow cytometry; The proportion of volunteers with binding antibody responses; All immune responses will be evaluated for proportion of responders and the mean responses will be compared.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Schlesinger, MD, Principal Investigator — The Rockefeller University
Locations (1):
- Rockefeller University, New York, New York, United States

REFERENCES:
- See also: Rockefeller Univesity research program information page — http://rucares.org